CLINICAL TRIAL: NCT01580761
Title: Sleep Restriction and Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Virend Somers, MD, PhD, MD, PhD, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 11-007272
Record Dates: First submitted 2012-04-17; First posted 2012-04-19 (Estimated); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sleep restriction (Experimental): Sleep restriction
  Interventions: Behavioral: Sleep restriction
- Normal sleep (No Intervention): Normal sleep

INTERVENTIONS:
Behavioral: Sleep restriction — 14 days of sleep restriction, 4 hours of sleep per day.
  Arms: Sleep restriction

SUMMARY:
Insufficient sleep may be one of the most common, and most preventable, obesity risk factors. The investigators wish to determine whether 14 nights of modest sleep restriction results in increased energy balance, thus potentially increasing the risk of obesity. The investigators hypothesize that sleep restriction will result in increased energy balance.

DETAILED DESCRIPTION:
Numerous studies have reported that self-reported short sleep duration is associated with obesity and weight gain. Insufficient sleep may be one of the most common, and most preventable, obesity risk factors. Given that sleep restriction is largely voluntary and potentially correctable, understanding the mechanisms that link insufficient sleep to positive energy balance and the development of obesity, particularly visceral obesity, is crucial to clinical applications, public health policy, and informing future studies. The investigators wish to determine whether 14 nights of modest sleep restriction results in increased energy balance, thus potentially increasing the risk of obesity. The investigators will combine energy balance, biomarker, and imaging data with state-of-the art sleep monitoring to provide unambiguous data on the effects of sleep restriction on obesity. Together, the investigators findings will help explain whether the reduced sleep duration in the general population may be contributing to the current epidemic of obesity, and suggest strategies to reduce this risk.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years
* BMI of 18.5-30 kg/m2
* Not a current smoker or tobacco user
* No chronic medical or psychiatric disorders
* On no prescription medications other than second generation antihistamines (cetirizine, fexofenadine, desloratadine, loratadine, etc), oral contraceptive pills, or intrauterine devices
* History of normal sleep patterns, defined as nocturnal sleep duration of 6.5-8 hours per night without regular daytime naps

Exclusion Criteria:

* The investigators will exclude subjects who have any medical or psychiatric disorders
* History of anxiety or depression
* Those taking any medications other than non-sedating antihistamines or oral contraceptives will be excluded
* Those found to have depression on a depression screening tool (BDI-II) will be excluded
* Current smokers will be excluded
* All female subjects will undergoing a screening pregnancy test and excluded if positive
* Subjects found to have significant sleep disorders will be excluded

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2012-07; Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Change in caloric intake and hunger | baseline to 21 days
  Change in caloric intake and hunger, measured during acclimation, experimental and recovery timepoints.
Change in energy expenditure | baseline to 21 days
  Change in energy expenditure, including activity energy expenditure, thermic effect of food (TEF), and basal metabolic rate (BMR), measured during acclimation, experimental and recovery timepoints..
Change in fat tissue characteristics and body composition | baseline to 21 days
  Changes in fat tissue characteristics from serial fat biopsies, and in body composition from DEXA and CT imaging, measured during acclimation, experimental and recovery timepoints.
Change in metabolic hormones | baseline to 21 days
  Change in metabolic hormones measured during acclimation, experimental and recovery timepoints.

SECONDARY OUTCOMES:
Change in neurocognitive deficits | baseline to 21 days
  Change in neurocognitive function measured by battery, measured during acclimation, experimental and recovery timepoints..
Change in blood pressure and autonomic function | baseline to 21 days
  Change in mean arterial blood pressure and autonomic function, measured during acclimation, experimental and recovery timepoints.
Change in markers of inflammation and endothelial function | baseline to 21 days
  Change in markers of inflammation and endothelial function, measured during acclimation, experimental and recovery timepoints.
Change in electrocardiographic characteristics | baseline to 21 days
  Change in electrocardiographic characteristics, measured during acclimation, experimental and recovery timepoints.
Change in arterial stiffness | baseline to 21 days
  Change in arterial stiffness, measured during acclimation, experimental, and recovery timepoints.
Change in cardiovascular reactivity | baseline to 21 days
  Change in cardiovascular reactivity, measured during acclimation, experimental, and recovery timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Virend Somers, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Covassin N, Singh P, McCrady-Spitzer SK, St Louis EK, Calvin AD, Levine JA, Somers VK. Effects of Experimental Sleep Restriction on Energy Intake, Energy Expenditure, and Visceral Obesity. J Am Coll Cardiol. 2022 Apr 5;79(13):1254-1265. doi: 10.1016/j.jacc.2022.01.038. PMID 35361348
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials